CLINICAL TRIAL: NCT01605240
Title: Ibuprofen vs. Codeine. Is One Better for Post-operative Pain Relief Following Reduction of Paediatric Forearm Fractures?
Brief Title: Ibuprofen Versus Codeine. Is One Better for Post-operative Pain Relief Following Reduction of Paediatric Forearm Fractures?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H2012:092
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Fracture; Pain
Keywords: Fracture pain; Fracture reduction; Analgesia; Acetaminophen; Ibuprofen; Codeine; Pediatric; Fracture Pain Analgesia in Pediatric population
MeSH Terms: conditions — Fractures, Bone; Pain; Agnosia | interventions — Acetaminophen; Ibuprofen; acetaminophen, codeine drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetaminophen and Codeine (Active Comparator): After their fracture is reduced, these patients will receive acetaminophen (15mg/kg) and codeine (1mg/kg) at regular dosing intervals.
  Interventions: Drug: Acetaminophen and Codeine
- Acetaminophen and Ibuprofen (Active Comparator): Following reduction of their fracture, these patients will receive acetaminophen (15mg/ml) and ibuprofen (10mg/ml) at regular dosing intervals.
  Interventions: Drug: Acetaminophen and Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen and Ibuprofen — After their fracture is reduced, these patients will receive acetaminophen (15mg/kg) and ibuprofen (10mg/kg) at regular dosing intervals.
  Other Names: Ibuprofen (Advil)
  Arms: Acetaminophen and Ibuprofen
Drug: Acetaminophen and Codeine — After their fracture is reduced, these patients will receive acetaminophen (15mg/kg) and codeine (1mg/kg) at regular dosing intervals.
  Arms: Acetaminophen and Codeine

SUMMARY:
For simple fractures treated in the emergency department with cast immobilisation only, ibuprofen has been shown to be superior to, or a least or equivalent to codeine with less side effects. These and other studies have commented that their results may not be applicable to children who have fractures that require reduction. There is currently no literature on the management of postoperative pain following reduction of paediatric fractures. The investigators aim therefore is to investigate whether either of the two most commonly prescribed analgesics is superior to the other for postoperative pain management following closed reductions of paediatric forearm fractures. Also, if one agent has more side effects than the other.

DETAILED DESCRIPTION:
This will be a prospective randomised controlled trial with the null hypothesis that there is no difference between ibuprofen and codeine in terms of pain relief or side effects.

Following ethics approval (submitted and approved) by the University of Manitoba ethics board a study group of fifty patients (25 in each arm) will be recruited to participate in the study.All patients will complete informed consent following both a verbal and written explanation of the study. Following the closed reduction they will all receive regular acetaminophen; (dose 15mg/kg) and either ibuprofen (10mg/kg) or codeine (1mg/kg) depending upon the group they were randomised to. This will have to be single blinding as the codeine formulation used by the hospital is a clear red liquid (5mg/ml) and the ibuprofen a cloudy colourless liquid (20mg/ml). They will also be given a "rescue" medication to be taken if the caregivers feel that the pain relief is not sufficient 1 hour after the study medication. This rescue medication will be the alternative medication in the study.

ELIGIBILITY:
Inclusion Criteria:

* All paediatric patients presenting to the section of paediatric orthopaedics requiring a closed reduction of a forearm fraction under either sedation or general anaesthetic.
* Patients who are able to return to follow up.

Exclusion Criteria:

* Any children with a history of gastrointestinal bleeding or ulceration, a bleeding disorder, a history of a low platelet count, a history of kidney disease, an uncontrolled chronic disease, or regular use of or allergy to acetaminophen, ibuprofen, or codeine.
* Children are also ineligible if they or their parents are unable to understand the consent process.
* Any child requiring anything other than a cast to supplement the stability of the fracture or an open reduction and internal fixation of the fracture.

Open fractures.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Pain Diary | Two Weeks
  Caregivers, or the children if old enough, will be asked to keep a pain diary. This will consist of the times the analgesia was taken and a pain score at awakening, at bedtime and before and 1 hour after each dose of medication.
  Caregivers/children will also be asked to include any side effects noted to medication and whether play, school, sleep, and eating are affected by pain each day. Caregivers will record whether the function was increased, decreased, or unchanged.

SECONDARY OUTCOMES:
Patient Satisfaction | 2 weeks
  Parent satisfaction will be measured each day with the use of a Likert 0-5 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Center, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Drendel AL, Lyon R, Bergholte J, Kim MK. Outpatient pediatric pain management practices for fractures. Pediatr Emerg Care. 2006 Feb;22(2):94-9. doi: 10.1097/01.pec.0000199564.64264.f4. PMID 16481924
- [Background] Drendel AL, Gorelick MH, Weisman SJ, Lyon R, Brousseau DC, Kim MK. A randomized clinical trial of ibuprofen versus acetaminophen with codeine for acute pediatric arm fracture pain. Ann Emerg Med. 2009 Oct;54(4):553-60. doi: 10.1016/j.annemergmed.2009.06.005. Epub 2009 Aug 19. PMID 19692147
- [Background] Koller DM, Myers AB, Lorenz D, Godambe SA. Effectiveness of oxycodone, ibuprofen, or the combination in the initial management of orthopedic injury-related pain in children. Pediatr Emerg Care. 2007 Sep;23(9):627-33. doi: 10.1097/PEC.0b013e31814a6a39. PMID 17876251
- [Background] Oakley EA, Ooi KS, Barnett PL. A randomized controlled trial of 2 methods of immobilizing torus fractures of the distal forearm. Pediatr Emerg Care. 2008 Feb;24(2):65-70. doi: 10.1097/PEC.0b013e318163db13. PMID 18277840
- [Background] Plint AC, Perry JJ, Correll R, Gaboury I, Lawton L. A randomized, controlled trial of removable splinting versus casting for wrist buckle fractures in children. Pediatrics. 2006 Mar;117(3):691-7. doi: 10.1542/peds.2005-0801. PMID 16510648
- [Background] Heidrich G, Slavic-Svircev V, Kaiko RF. Efficacy and quality of ibuprofen and acetaminophen plus codeine analgesia. Pain. 1985 Aug;22(4):385-397. doi: 10.1016/0304-3959(85)90044-2. PMID 4047707
- [Background] Clark E, Plint AC, Correll R, Gaboury I, Passi B. A randomized, controlled trial of acetaminophen, ibuprofen, and codeine for acute pain relief in children with musculoskeletal trauma. Pediatrics. 2007 Mar;119(3):460-7. doi: 10.1542/peds.2006-1347. PMID 17332198
- [Background] Bieri D, Reeve RA, Champion DG, Addicoat L, Ziegler JB. The Faces Pain Scale for the self-assessment of the severity of pain experienced by children: development, initial validation, and preliminary investigation for ratio scale properties. Pain. 1990 May;41(2):139-150. doi: 10.1016/0304-3959(90)90018-9. PMID 2367140